CLINICAL TRIAL: NCT04031482
Title: TARGET Registry A Project of the German Network for Intestinal Diseases in Cooperation With the German Association of Gastroenterologists in Private Practice (Bng) and Other Corporate Partners
Brief Title: TARGET Registry A Project of the German Network for Intestinal Diseases in Cooperation With Other Corporate Partners
Acronym: TARGET
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ced Service GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1.2
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Crohn Disease; Ulcerative Colitis; Indeterminate Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ongoing or incipient targeted therapies: Ongoing or incipient targeted therapies with biologics and/or other targeted therapies (e.g. Janus kinase inhibitors)
  Interventions: Other: No intervention, only standard care

INTERVENTIONS:
Other: No intervention, only standard care — The aim of this registry is to expand on previous findings in the field of diagnostic and therapeutic pathways for patients with Crohn's disease, ulcerative colitis and indeterminate colitis undergoing routine administration of a targeted therapy (biologics or another targeted therapy such as Janus kinase therapy) and various different treatment approaches. A data pool is to be generated for this purpose, in order to
  * analyse disease progression
  * systematize findings about treatment processes
  * identify potential influencing factors
  * review any new diagnostic procedures
  * identify potential test subjects for further study
  * evaluate the safety of various treatment concepts

SUMMARY:
By capturing possible or known risk factors, it will be possible to recognize connections between these risk factors and the disease, thus obtaining valuable insights into the cause of the disease. This in turn facilitates an improved evaluation of the treatment situation as well as influencing future framework conditions for preventive measures and planning treatments. Disease registries are thus crucial for the planning and structuring of health policies.

The present registry protocol serves as a basis for the proper implementation of a registry for patients with chronic inflammatory bowel diseases. It describes the study rationale, objectives, design, participant groups, procedures and evaluation methods. Furthermore, it defines the responsibilities of each person involved in maintaining the registry and also forms the basis for decisions regarding evaluation by the Ethics Committee.

DETAILED DESCRIPTION:
In view of the high prevalence and currently unsatisfactory treatment status, there is a significant medical demand for more effective treatment options. These require greater knowledge about the condition in the form of full disease progressions while exposed to a wide range of different treatment concepts and influencing factors. It has been possible to significantly increase scientific understanding of the pathogenesis of ulcerative colitis and Crohn's disease over the last few decades. Clinical and experimental results indicate a causal link with gastrointestinal barrier dysfunction and defective regulation of the immune system. However, no evidence has been found to prove that patients with the disease develop an immune deficiency by themselves, resulting in an increased susceptibility to bacterial or viral infections. Furthermore, there are unanswered questions concerning aetiology, risk factors and influencing factors for the early prediction of treatment responses.

The aim of this registry is to expand on previous findings in the field of diagnostic and therapeutic pathways for patients with Crohn's disease, ulcerative colitis and indeterminate colitis undergoing routine administration of a targeted therapy (biologics or another targeted therapy such as Janus kinase therapy) and various different treatment approaches. A data pool is to be generated for this purpose, in order to

* analyse disease progression
* systematize findings about treatment processes
* identify potential influencing factors
* review any new diagnostic procedures
* identify potential test subjects for further study
* evaluate the safety of various treatment concepts

A specific objective has not been defined for this registry as a registry does not per se need to build upon the foundation of a theoretically-deduced research hypothesis. Rather, it acts as a gateway for generating a systematic data repository.

The registry offers researchers the opportunity to formulate their own research hypotheses based on the collected data and to then use the generated data pool to attempt to test their hypothesis. Additional data/variables could also be collected as necessary in order to answer certain questions.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Crohn's disease or Confirmed diagnosis of ulcerative colitis or Confirmed diagnosis of indeterminate colitis (IBDU)
2. All types of treatment commensurate with the medical practice, independent of any study
3. Age 18-80
4. Ongoing or incipient targeted therapies with biologics and/or other targeted therapies (e.g. Janus kinase inhibitors)
5. Sufficient ability to communicate in German language
6. Patient must be able to recognize the nature, significance and scope of this registry and to act accordingly
7. Computer/Tablet/mobile phone with internet access

Exclusion Criteria:

1. No declaration of consent is given
2. Age < 18 and > 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with a confirmed diagnosis of Crohn's disease, ulcerative colitis or indeterminate colitis who is undergoing a targeted therapy is a potential candidate for taking part in the registry.
Sampling Method: Probability Sample
Enrollment: 4400 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Disease activity | 3 Years
  harvey bradshaw index

OTHER OUTCOMES:
Quality of life (QOL) | 3 Years
  The Questioner EQ-5D is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D expresses the state of health of the respondents in a one-dimensional measure from 0 (very poor) to 1 (best possible state of health).
Use of glucocorticoids | 3 Years
  Use of glucocorticoids
Need for surgery | 3 Years
  Need for surgery
Occurrence of side effects and infections | 3 Years
  Occurrence of side effects and infections
Longevity of started treatments | 3 Years
  Longevity of started treatments

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Plachta-Danielzik, PD Dr., Study Director — Kompetenznetz Darmerkrankungen

IPD SHARING:
Plan to Share IPD: Undecided